CLINICAL TRIAL: NCT00434070
Title: Comparison of the Development of Thymidine Analogue Mutations With CD4 Monitoring Alone Versus CD4 Monitoring Plus Viral Load Monitoring in Naive HIV-1 Individuals on First-Line Antiretroviral Therapy in Africa
Brief Title: Relationship of Viral Resistance Development to CD4 Monitoring Alone or With Viral Load Monitoring
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907093; 07-I-N093
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2013-02-07

CONDITIONS: Acquired Immunodeficiency Syndrome; Resistance
Keywords: HIV; Antiretrovial Therapy; Resistance; Monitoring; TAMS; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine whether HIV-infected patients are more likely to develop resistance to antiretroviral therapy if their blood is not monitored for the number of viruses (viral load) in the body.

A virus that changes (mutates) over time may become resistant to certain types of medicine. This resistance may affect future treatment options. This study will compare the amount of virus in the blood of HIV-infected patients who have been monitored for viral load with the amount of virus in the blood of patients who have not been monitored for viral load. For patients who have detectable virus, the type of resistance (mutations) of the virus will be determined by comparing the components of the virus with that of a virus that is known not to be resistant.

HIV-infected patients 18 years of age or older who are being treated at the Infectious Diseases Institute at Mulago Hospital at Makerere University in Kampala, Uganda, may be eligible for this study. Participants are interviewed about the treatments they have received for HIV and how they usually take their anti-HIV drugs. They also have a blood sample drawn for research tests.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) has become widely available in resource limited settings (RLS) due to large increases in available resources through the President s Emergency Plan for AIDS Relief (PEPFAR) and the Global Fund for AIDS, Tuberculosis, and Malaria (GFATM). The number of people accessing ART in RLS doubled in 2005 alone. Whereas viral load testing is done routinely for individuals on ART in the western hemisphere, this is not the case elsewhere. The World Health Organization (WHO) has recommended only clinical and CD4 count monitoring as the standard of care in RLS during the ART scale-up. As a result, there is a growing population of individuals in Africa currently on ART whose treatment is monitored only using clinical evaluations and CD4 counts.

In addition to preserving lives and improving the quality of life of HIV infected individuals, the goal of ART is to achieve and maintain suppression of HIV replication to an undetectable level. This goal enables the treatment to remain effective in the long term since the emergence of resistant strains is limited by the low replication rate of HIV achieved under these conditions. The recovery of the immune system as determined through CD4 count monitoring is neither a very sensitive nor specific marker of virological suppression in individuals on ART. Therefore, monitoring the response to ART using just the WHO guidelines for RLS may lead to a significant delay in detecting the failure to achieve or maintain virological suppression among individuals who are failing treatment. This is in contrast to western settings where routine viral load testing leads to early detection of failure to achieve suppression.

Failure to monitor and detect unsuppressed virus increases the risk of development of resistance to ART. In particular, failure to achieve or maintain virologic suppression for prolonged periods of time may lead to the sequential development of thymidine analogue mutations (TAMs) in patients taking zidovudine (AZT) or stavudine (d4T) as part of ART regimens. The accumulation of 3 or 4 TAMs confers drug resistance across the nucleoside reverse transcriptase inhibitors (NRTI) class of antiretroviral (ARV) drugs and has implications for future ART regimens, particularly in RLS where second line ART options are limited. Stavudine and zidovudine are currently used as part of the first line regimens in Sub-Saharan Africa and other RLS areas.

We hypothesize that patients who are monitored with a combination of CD4 counts and viral load measurements routinely develop TAMs at a slower rate than do patients who are monitored with only CD4 count measurement (as per WHO guidelines in RLS). This hypothesis is based on the higher risk of delay in detection of unsuppressed virus in patients who are monitored by clinical and CD4 counts alone, which may translate into the development of drug-resistant mutations.

The study team therefore proposes to carry out a cross-sectional study in a large public HIV out-patient clinic in which patients who are routinely monitored with both CD4 count and viral load measurements are compared with patients who are routinely monitored with CD4 counts measurement only. Individuals who have detectable viral load after 36 months of ARV therapy in each of the above patient categories shall undergo a structured interview and HIV genotypic testing, particularly to look for TAMs. The presence of TAMs in each instance shall be documented.

The results of this study will highlight the magnitude of the risk of using CD4 count monitoring only in patients on ART in RLS and contribute to efforts to find cheaper technologies for virological monitoring of these individuals. The findings will also support the choice of second line drug regimens that may be proposed for use in Africa.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Willing to provide individual informed consent.
  2. HIV positive. (HIV status will have been confirmed by recognized external testing centre (e.g., AIC) or if necessary by the IDI lab using Abbott Determine HIV1-2 plus STAT-PAK (Chembio Diagnostic Systems) rapid tests. Unigold (Trinity Biotech) is available for tie-breaker testing if necessary.
  3. Currently being followed at the Adult Infectious Disease Clinic.
  4. Patients who are aged 18 years or more.
  5. Patients who initiated ART therapy at the Adult Infectious Disease Clinic (First line ART regimens include either stavudine or zidovudine).
  6. Patients who were ART naive at ART initiation (from patient medical record).
  7. Patients who have been on ART for at least 36 months and no greater than 40 months.

EXCLUSION CRITERIA:

1. Inability or unwillingness to provide individual informed consent.
2. Patients currently admitted to Urgent Care facility (severely ill).
3. Age less than 18 years.
4. Presence of a documented infection within a period of 4 weeks from screening for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2007-02-07; Study Completion 2013-02-07

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

REFERENCES:
- [Background] Akileswaran C, Lurie MN, Flanigan TP, Mayer KH. Lessons learned from use of highly active antiretroviral therapy in Africa. Clin Infect Dis. 2005 Aug 1;41(3):376-85. doi: 10.1086/431482. Epub 2005 Jun 30. PMID 16007536
- [Background] Deeks SG, Grant RM. Sustained CD4 responses after virological failure of protease inhibitor-containing therapy. Antivir Ther. 1999;4 Suppl 3:7-11. PMID 16021865
- [Background] Weiss L, Burgard M, Cahen YD, Chaix ML, Laureillard D, Gilquin J, Piketty C, Viard JP, Kazatchkine MD, Girard PM, Rouzioux C. Immunological and virological features of HIV-infected patients with increasing CD4 cell numbers despite virological failure during protease inhibitor-based therapy. HIV Med. 2002 Jan;3(1):12-20. doi: 10.1046/j.1464-2662.2001.00095.x. PMID 12059946